CLINICAL TRIAL: NCT02706379
Title: The Impact of Early Goal-Directed Therapy to Perfusion and Metabolism of Brain in Septic Shock Patients
Brief Title: Impact of Early Goal-Directed Therapy to Perfusion and Metabolism of Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, director, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015ZDSYLL036.0
Record Dates: First submitted 2015-12-11; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Local cerebral oxygen saturation (Experimental): use NIRS technical to detect local cerebral oxygen saturation of both sides of brain
  Interventions: Other: Local cerebral oxygen saturation

INTERVENTIONS:
Other: Local cerebral oxygen saturation — take blood culture before antibiotic use;measure the blood lactate;liquid rescisutation as 20ml/kg

SUMMARY:
Early goal directed therapy (EGDT) is an effective treatment for patients with septic shock, which is widely used in clinic. Fluid resuscitation can significantly reduce the mortality of patients with septic shock and improve the prognosis of patients with EGDT. However, in recent years, the standard of EGDT to determine the existence of the target of septic shock. Some studies have shown that there may be a manifestation of the deficiency of kidney and liver and other organs such as kidney, liver and other organs in the recovery of EGDT. Therefore, this experiment is to explore the brain perfusion and metabolism of the EGDT when the target is reached.The aim of this study was to investigate the effects of EGDT as a guide to the cerebral perfusion and metabolism in order to provide clinical evidence for the treatment of fluid resuscitation in patients with septic shock.

DETAILED DESCRIPTION:
1. patients enrollment this project: Met the inclusion criteria without exclusion criteria were entered test, and record the general information, including name, hospital number, gender, age, height, weight, admission, and in time, ICU admission and in ICU diagnosis, previous underlying diseases, into the group of APACHE II score and SOFA score
2. implement septic shock bundle: measurement the value of lactic acid of patients after administrating of ICU, take blood culture before antibiotic using, give wide-spectrum antibiotic treatment and began liquid resuscitation
3. preparation： A. basic state records B. using CAM-ICU delirium assessment for patients, and record the assessment results C. cerebral oxygen saturation monitor D. via the jugular vein placed central venous catheter and femoral artery placed PiCCO catheter
4. monitoring of hemodynamics and cerebral perfusion and metabolic indicators

ELIGIBILITY:
Inclusion Criteria:

* New infectious shock in accordance with the diagnostic criteria of the 2012 SSC guidelines；
* Liquid recovery is not fully achieved EGDT standards, at least meet the following criteria:

  * mean arterial pressure < 65mmHg
  * central venous pressure < 8mmHg
  * per hour urine volume was less than 0.5ml/kg
  * central venous oxygen saturation <70%
  * arterial blood lactic acid value > 2.5mmol/L
* Signed informed consent

Exclusion Criteria:

* Subjects/subjects client reject the invasive hemodynamic monitoring
* have contraindications to place hemodynamic monitoring
* unconsciousness state before septic shock and GCS<12
* cannot put the electrodes on the eyebrow
* pregnant or lactating women
* end stage of illness or death rate is more than 80%

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
change of local cerebral oxygen saturation between early goal directed treatment(EGDT) | through study completion, up to 6 hours
  Test the local cerebral oxygen saturation of both sides of brain through near infrared spectroscopy technology. And record the change of local cerebral oxygen of the left and right's brain.

SECONDARY OUTCOMES:
change of neuron specific enolase(NSE) | through study completion, up to 6 hours
  NSE is an enzyme that in humans is encoded by the ENO2 gene. NSE is produced by small cell carcinomas which are neuroendocrine in origin, and the raise of its concentration indicates the injury of brain.
change of S-100 protein | through study completion, up to 6 hours
  S-100 protein S100 proteins are normally present in cells derived from the neural crest (Schwann cells, and melanocytes), chondrocytes, adipocytes, myoepithelial cells, macrophages, Langerhans cells, dendritic cells, and keratinocytes.S100 proteins have been implicated in a variety of intracellular and extracellular functions.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Doctor, Study Director — 13951965301

IPD SHARING:
Plan to Share IPD: No
The data is personal, and will not share to others.